CLINICAL TRIAL: NCT00106093
Title: Assessment and Treatment of People With Alcohol Drinking Problems
Brief Title: Alcoholism Assessment and Treatment
Status: Completed | Type: Observational
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050121; 05-AA-0121
Record Dates: First submitted 2005-03-19; First posted 2005-03-21 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2015-09-08

CONDITIONS: Alcoholism; Alcohol Dependence; Alcohol Drinking Related Problems
Keywords: Alcohol; Alcohol Treatment; DNA; Treatment; Alcohol Dependence; Alcoholism; Alcohol Drinking Related Problems
MeSH Terms: conditions — Alcoholism

SUMMARY:
The purpose of this study is to gather information about people s drinking histories and to evaluate them for other research studies being conducted at the National Institute on Alcohol Abuse and Alcoholism (NIAAA). The evaluation will include a physical examination, blood tests, an MRI scan of the brain and completion of various questionnaires about alcohol use and mood. The information gathered from all of these tests will be used by researchers to gain a better understanding of the disease of alcoholism and determine eligibility for other NIAAA studies. This is an inpatient study so participants will stay at the NIH hospital for at least three weeks and up to six weeks if a person is found to be eligible for other NIAAA research studies.

The study is open to people age 18 and older whose alcohol drinking has caused significant problems in their lives, and who desire alcoholism treatment. Detoxification will be provided if needed, and each person may participate in our alcoholism treatment program. The treatment includes group and individual counseling sessions as well as self-help meetings such as AA. Family counseling and recreational opportunities are also an important part of the treatment experience. The doctors, nurses, social workers and all of our other staff are committed to helping participants design an aftercare program that will help them leave the hospital and remain sober. Participants may also be able to attend a 12-week aftercare program in the NIAAA outpatient clinic.

DETAILED DESCRIPTION:
OBJECTIVE: The purpose of this protocol is to create a mechanism whereby the intramural program of the NIAAA can evaluate and treat a broad range of people with drinking problems at the NIH Clinical Center (CC) in Bethesda, MD. Through this program, participants will receive comprehensive, state-of-the-art treatment for their alcohol, psychosocial and medical problems. The protocol will allow us to evaluate and recruit participants who will then be eligible for more focused clinical research efforts to advance the NIAAA research goals. Additionally, this protocol will allow investigators and staff to gain broad training experience in alcohol and addiction medicine through the clinical care of such patients.

STUDY POPULATION: The protocol is open to any adult who is seeking help for a drinking problem and who is likely to qualify to participate in another NIAAA protocol. Participants will be recruited through local media and professional avenues in the Washington, DC Metro area.

DESIGN: Participants will be evaluated by a nurse and physician, among others, who will determine the need for hospitalization, detoxification and to address other issues. For those needing medically supervised detoxification, a standard program of monitoring and treatment with benzodiazepines and other medications will be instituted. A standard battery of screening blood, urine and other clinically indicated tests, an electrocardiogram, chest x-ray and MRI of the brain will be done as part of the comprehensive medical and

neurological assessment. Following admission, participants will undergo a series of verbal and observational-type assessments designed to evaluate psychiatric co-morbidity, psychopathology, psychosocial problems, neurocognitive function, personality and other factors relevant to alcoholism treatment. Following discharge from the inpatient program, participants will be offered up to 16 weeks standard-of-care behavioral outpatient treatment. At five points during the outpatient phase, participants will come to the clinic for selected blood and urine tests, interviews and verbal/observational assessments to evaluate abstinence from alcohol and identify changes in various psychological dimensions. During their participation in this protocol, participants will be approached to consider enrolling in other clinical research protocols such as imaging studies and drug-treatment trials. For participants willing to participate in these other protocols, other appropriate consent(s) will be obtained.

OUTCOME MEASURES: Because of the evidence-based nature of all assessments used in this protocol, data obtained through them can serve at least three clinical purposes: first, to provide a basis for individualizing patient treatment, enhancing motivation to change, and following-up such treatment for the sole purpose of providing optimal clinical care; second, to provide patient characteristics and outcome data for specific research protocols to which the patient may additionally and separately consent; and third, to provide data for monitoring the performance and functioning of the program as a whole.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age greater than 18 years old.

Are seeking help for alcohol drinking-related problems.

EXCLUSION CRITERIA:

People with medical problems that cannot be adequately managed at the NIH Clinical Center, as determined by the medically advisory investigator, in consultation with relevant Clinical Center consult services as needed.

Serious neuro-psychiatric conditions which impair judgment or cognitive function to an extent that precludes them from providing informed consent, such as acute psychosis or severe dementia (incompetent individuals).

People who are unlikely or unable to complete the treatment program because they become or are likely to be incarcerated while on the protocol.

People who are required to receive treatment by a court of law or who are involuntarily committed to treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1192 (Actual)
Dates: Start 2005-03-16; Study Completion 2015-09-08

CONTACTS AND LOCATIONS:
Overall Officials: Nancy DiazGranados, M.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] O'Connor PG, Schottenfeld RS. Patients with alcohol problems. N Engl J Med. 1998 Feb 26;338(9):592-602. doi: 10.1056/NEJM199802263380907. No abstract available. PMID 9475768
- [Background] COMBINE Study Research Group. Testing combined pharmacotherapies and behavioral interventions in alcohol dependence: rationale and methods. Alcohol Clin Exp Res. 2003 Jul;27(7):1107-22. doi: 10.1097/00000374-200307000-00011. PMID 12878917
- [Background] O'Brien CP. Treatment of alcoholism as a chronic disorder. Alcohol. 1994 Nov-Dec;11(6):433-7. doi: 10.1016/0741-8329(94)90063-9. PMID 7865139
- [Derived] Wallen GR, Brooks AT, Whiting B, Clark R, Krumlauf MC, Yang L, Schwandt ML, George DT, Ramchandani VA. The prevalence of sleep disturbance in alcoholics admitted for treatment: a target for chronic disease management. Fam Community Health. 2014 Oct-Dec;37(4):288-97. doi: 10.1097/FCH.0000000000000040. PMID 25167069